CLINICAL TRIAL: NCT06567444
Title: Improving Cognitive Function in Chinese Children With ADHD and/or RD Through Computerized Working Memory Training
Brief Title: Computerized Working Memory Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EdUHK_WM
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: ADHD; Dyslexia
Keywords: ADHD; dyslexia; executive function; intervention; training app; working memory
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dyslexia

STUDY DESIGN:
Intervention Model Description: A single-blind study design was adopted in which all assessors were blinded to the treatment condition of the students. There were three experimental groups, with 26 participants in the ADHD group, 38 participants in the RD group, and 24 participants in the ADHD+RD group. The typically developing control group had 32 participants.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ADHD Group (Experimental): This experimental group received the working memory training conducted in primary schools in Hong Kong. This group was led by trained research assistants.
  Interventions: Other: Working memory intervention
- RD Group (Experimental): This experimental group received the working memory training conducted in primary schools in Hong Kong. This group was led by trained research assistants.
  Interventions: Other: Working memory intervention
- ADHD+RD Group (Experimental): This experimental group received the working memory training conducted in primary schools in Hong Kong. This group was led by trained research assistants.
  Interventions: Other: Working memory intervention
- TD Group (No Intervention): The participants in the TD group did not receive any training.

INTERVENTIONS:
Other: Working memory intervention — During the intervention, the participants in the ADHD group received five computerized working memory training sessions per week over five weeks, and each session lasted 20 minutes. This training paradigm is based on previous studies which show improvements in working memory capacities after a 5-week training period.
  Arms: ADHD Group; ADHD+RD Group; RD Group

SUMMARY:
Prior research has found that children with attention-deficit hyperactivity disorder (ADHD) and reading difficulties (RD) are at an elevated risk of developing further cognitive deficits and developmental challenges. ADHD and RD are characterized by a deficit in working memory, which negatively affects learning and behavior. The main aims of this study were to design a working memory training app and examine its effectiveness through a 5-week training program in Chinese children with ADHD and/or RD. There were three experimental groups, with 26 participants in the ADHD group, 38 participants in the RD group, and 24 participants in the ADHD+RD group. The typically developing (TD) control group had 32 participants. All participants completed the pretest and posttest assessments on executive function and reading performance.

DETAILED DESCRIPTION:
Attention-deficit hyperactivity disorder (ADHD) is marked by attention issues and hyperactive-impulsive behaviors. It affects about 7.2% of school-aged children globally, with a 6.5% prevalence in Hong Kong. Reading difficulties (RD) involve persistent challenges in reading and writing, unrelated to brain damage, sensory impairments, or low intelligence. ADHD and RD often co-occur, with a comorbidity rate of 25%-40%, surpassing chance probabilities.

Research indicates that children facing the dual challenge of ADHD and RD are more vulnerable to significant cognitive deficits, particularly in working memory. This vital cognitive function strongly influences academic abilities like math problem-solving, reading, and language understanding. Deficiencies in working memory can result in learning overwhelm, memory lapses with instructions, and struggles with complex tasks in children. Consequently, individuals with this comorbidity are predisposed to more challenges compared to those with a singular disorder.

Studies have verified that individuals with both ADHD and RD symptoms face increased chances of school abandonment, disruptive conduct, delinquency, and notably, more aggression compared to those with singular conditions. These results emphasize the need for additional research to develop a fresh intervention strategy targeting this comorbid cohort, aiming to pre-empt these adverse consequences. The subsequent sections will provide a concise overview of the theoretical basis of working memory and its ties to ADHD and RD, followed by the development of a working memory training application and the research methodology.

Working memory, a crucial cognitive function, involves temporarily storing, processing, and recalling information within specific limits. It underpins various mental processes like problem-solving, language comprehension, and fluid intelligence. This ability is vital for learning new concepts and skills, correlating strongly with vocabulary growth, language understanding, and reading ability. Baddeley and Hitch's influential working memory model includes a central executive, the phonological loop, the visuospatial sketchpad, and later, the episodic buffer. The central executive plays a pivotal role in coordinating these components, managing data retrieval and manipulation while allocating resources to the storage systems.

The phonological loop specializes in processing language-related data crucial for language learning. Meanwhile, the visuospatial sketchpad handles visual and spatial information, linked to nonverbal intelligence and orthographic awareness. The episodic buffer acts as a unified episodic representation, capable of integrating data from other components and long-term memory. This model illuminates how working memory functions, influences cognitive processes, and develops over time.

Working memory is vital for various cognitive functions, with its components showing distinct links to ADHD and RD. Notably, ADHD often presents with noticeable working memory deficits, underscoring its significance in the cognitive makeup of individuals with ADHD. The response inhibition model of ADHD suggests that deficient response inhibition is a core issue leading to executive function problems, including working memory challenges. The central executive element, along with subsystems like the phonological loop and visuospatial sketchpad, plays critical roles in this context. Deficiencies in the central executive are thought to manifest as key ADHD symptoms. While verbal working memory issues are consistently observed in ADHD, visuospatial working memory impairments may vary in severity, indicating a multifaceted working memory profile in ADHD, pivotal to the condition's cognitive characteristics.

RD is frequently linked with working memory deficiencies, particularly in the phonological realm. The phonological loop, a key working memory element responsible for temporarily managing and processing speech-based data, plays a crucial part in these shortcomings. Numerous studies consistently demonstrate that individuals with RD encounter difficulties in activities demanding effective phonological loop operation, like verbal memory span tasks. However, recent studies suggest that working memory impairments in dyslexia may transcend phonological processing. Emerging research indicates issues with the central executive aspect of working memory, indicating broader cognitive hurdles in individuals with RD. Challenges in visuospatial processing may also be present in individuals with RD, especially in tasks requiring verbal mediation, underscoring the intricate nature of working memory deficits in RD.

These findings underscore the critical importance of working memory in both ADHD and RD. In ADHD, deficits primarily affect the central executive function, impacting core aspects of working memory, whereas in RD, deficits in phonological processing within working memory are more prominent. While this deficiency is present in both standalone ADHD and RD groups, it appears more pronounced in individuals with comorbid conditions. Wang and Chung's study demonstrates that working memory effectively distinguishes Taiwanese children with comorbid ADHD and RD symptoms from those in singular-deficit groups (ADHD or RD alone) and typically developing children. Recent research by Poon and colleagues suggests that, compared to individual ADHD and RD groups, comorbid groups exhibit additional deficits in central executive function, a critical aspect involving information retention for task completion, which is not observed in singular groups. These results emphasize the importance of early intervention training for this specific group of children.

Over the last 15 years, there has been a significant increase in the use of medication for children with ADHD, with a 36-fold rise in Hong Kong and a 34-fold increase in the UK. In the United States, Danielson and colleagues found that 62% of children with ADHD are on medication. While pharmaceutical interventions can effectively help manage ADHD symptoms, they also come with potential side effects like insomnia, reduced appetite, mood swings, and stunted growth. Additionally, the long-term efficacy of such treatments may be limited, and symptoms could reappear once the medication is ceased. While pharmaceutical treatments have proven effective in addressing the core symptoms of ADHD, their applicability to comorbid conditions remains a subject of ongoing discussion.

Some studies indicate that pharmacological treatments, such as psychostimulants and non-stimulant medications, can effectively mitigate symptoms linked to ADHD, like inattention, hyperactivity, and impulsivity. These treatments are often seen as crucial in enhancing the daily functionality and well-being of children with ADHD. Nonetheless, it is important to recognize that the impact of pharmacological interventions on comorbid conditions can vary, and they may not consistently yield the same level of improvement across all areas. For example, while ADHD symptoms might respond positively to pharmacological treatments, the same level of efficacy may not be observed for comorbid reading difficulties, as suggested by some researchers.

The administration of psychostimulant medication in cases of comorbidity can yield varying outcomes depending on the specific conditions involved. Research suggests that some children with ADHD and comorbid RD may experience improvements in executive functioning, behavior, and reading abilities with medication. However, responses to medication are highly individualized, and not all children may benefit significantly. It is crucial to carefully consider the potential benefits against the risks and side effects, especially in cases of comorbidity. In the context of ADHD and comorbid conditions, the decision to use psychostimulants or other medications is complex and multifaceted. Factors such as individual needs, parental preferences, and the presence of contraindications all play a role in determining the appropriateness of medication use. It is essential for healthcare professionals to consider these factors and engage in thorough discussions with patients and caregivers to make informed decisions regarding treatment options.

The effectiveness of pharmacological treatments in cases of comorbid conditions remains a subject of continuous research and debate, underscoring the necessity for comprehensive, multimodal strategies to tackle the complex challenges faced by children with ADHD and RD. This study delves into one such approach-working memory training-and its potential to offer advantages to this specific group of children. Through an investigation into the efficacy of working memory training, the aim is to contribute to a deeper comprehension of interventions that could potentially bolster the cognitive and academic skills of these individuals. Such research could pave the way for more tailored and effective interventions that address the diverse needs of children dealing with both ADHD and RD.

Research has firmly established that working memory can be improved through training that targets the prefrontal cortical circuits. The brain's plasticity allows it to continuously adjust to its surroundings. Studies on neural systems have pinpointed "sensitive periods" when specific brain regions are highly responsive to environmental cues. Neuroimaging research demonstrates that changes in neural activation patterns resulting from computerized training often correspond to enhanced working memory capacity. These insights showcase the brain's adaptability and the promise of tailored interventions to boost cognitive functions such as working memory by engaging specific neural pathways effectively.

Computerized working memory training has proven effective in reducing ADHD symptoms and enhancing visual domains. Klingberg et al.'s five-week program notably boosted working memory capacity and behaviors in students with ADHD. Similarly, Luo et al. reported improvements in working memory, especially in visual tasks, for children with RD undergoing specific training. However, no training to date has integrated both storage pathways as proposed by Barkley's model. To address this gap, the first author developed an app combining phonological and visuo-spatial working memory training using n-back and card pairing exercises.

Children with ADHD and/or RD often face challenges due to poor working memory, leading to various developmental issues. The rise in ADHD and RD cases, along with increased medication usage, has drawn attention. Many educators and caregivers seek non-medication solutions to enhance cognitive function in these children. This study aims to assess the impact of computerized working memory training on different memory areas and reading skills in ADHD, RD, ADHD+RD, and typically developing groups. The goal is to introduce this new training app to assist teachers and parents in supporting children with ADHD and/or RD both at school and home.

ELIGIBILITY:
Inclusion Criteria:

* being aged between 6 and 11
* having an intelligence quotient (IQ) score above 80
* having a clinical diagnosis of ADHD and/or RD from a clinical or educational psychologist or a psychiatrist
* speaking native Cantonese

Exclusion Criteria:

* brain damage, neurological issues, sensory problems, or psychiatric issues

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Intellectual ability | Two weeks before the pretest
  The Raven's Progressive Matrices comprises five sets (starting with set A and ending with set E) of 12 items each, totalling 60 items. Each presents a visual pattern with a missing piece. Participants were required to identify the missing piece that would complete the pattern.
Central executive function | One week before the intervention
  The central executive function subscale of BRIEF consists of 10 items. Teachers rated their student's behavior using a 3-point Likert scale (1 = never, 2 = sometimes; 3 = often). All 10 items were added together to form the central executive function subscale.
Central executive function | One week after the intervention
  The central executive function subscale of BRIEF consists of 10 items. Teachers rated their student's behavior using a 3-point Likert scale (1 = never, 2 = sometimes; 3 = often). All 10 items were added together to form the central executive function subscale.
Verbal working memory | One week before the intervention
  Verbal working memory capacity was measured using the third edition of the backward digit spans subtest from the Wechsler Intelligence Scale for Children (WISC-III). Participants were presented with two to nine orally delivered digits and asked to recall them in reverse order. They must retain auditory information while filtering out irrelevant details and focusing on relevant ones. The backward digit spans subtest consists of 18 trials, and participants who correctly repeated the backward digit sequence received one point.
Verbal working memory | One week after the intervention
  Verbal working memory capacity was measured using the third edition of the backward digit spans subtest from the Wechsler Intelligence Scale for Children (WISC-III). Participants were presented with two to nine orally delivered digits and asked to recall them in reverse order. They must retain auditory information while filtering out irrelevant details and focusing on relevant ones. The backward digit spans subtest consists of 18 trials, and participants who correctly repeated the backward digit sequence received one point.
Visual-spatial working memory | One week before the intervention
  Visual-spatial working memory was assessed using the Spatial Working Memory Test (SWM) from Cambridge Cognition. This computerized measure presents several boxes on the screen. Participants were asked to locate a hidden yellow token in each search. Once the token is collected, participants must continue searching for the remaining tokens until all of them have been found (the number of tokens equals the number of boxes). The token never appears in boxes where one has been found before. The number of boxes increases in difficulty from four to eight.
Visual-spatial working memory | One week after the intervention
  Visual-spatial working memory was assessed using the Spatial Working Memory Test (SWM) from Cambridge Cognition. This computerized measure presents several boxes on the screen. Participants were asked to locate a hidden yellow token in each search. Once the token is collected, participants must continue searching for the remaining tokens until all of them have been found (the number of tokens equals the number of boxes). The token never appears in boxes where one has been found before. The number of boxes increases in difficulty from four to eight.
Chinese word reading | One week before the intervention
  The 1-minute word reading test from HKT-P(III) was used to measure reading fluency. It consists of 120 simple Chinese two-character words. Participants were asked to read the words as quickly and accurately as possible within a minute. The total number of words read correctly was recorded, and the reading ability score can vary between 0 and 120.
Chinese word reading | One week after the intervention
  The 1-minute word reading test from HKT-P(III) was used to measure reading fluency. It consists of 120 simple Chinese two-character words. Participants were asked to read the words as quickly and accurately as possible within a minute. The total number of words read correctly was recorded, and the reading ability score can vary between 0 and 120.

CONTACTS AND LOCATIONS:
Locations (1):
- The Education University of Hong Kong, Tai Po, Hong Kong

REFERENCES:
- [Derived] Poon K, Ho MSH, Wang LC, Lee HM, Lau WKW, Chan WWL. Improving cognitive function in Chinese children with ADHD and/or RD through computerized working memory training. BMC Psychol. 2024 Oct 18;12(1):574. doi: 10.1186/s40359-024-02065-1. PMID 39425120